CLINICAL TRIAL: NCT03946436
Title: Impact of Active Video Games on Motor- and Visual Spatial-learning Capabilities During the Process of Tennis Training in Young Children
Brief Title: Playing AVI During Tennis Training Process
Acronym: AVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marusic (Other)
Collaborators: Science and Research Centre Koper (Other); University of Primorska (Other)
Responsible Party: Sponsor-Investigator, Marusic, Assistant professor Uros Marusic, PhD, Science and Research Centre Koper
Organization: Science and Research Centre Koper (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVITENNIS
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Learning, Spatial; Cognitive Change
Keywords: stroke technique; psychophysiological body responses; visual perceptual skills; reaction time.
MeSH Terms: conditions — Spatial Learning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-AVI (Experimental): The I-AVI group were involved in a regular tennis training process, two times a week for one hour. Additionally right after the tennis lessons they played a Virtua Tennis 4 active video game for 20 minutes per participant. They use the playstation kinect console. The intervention lasted 6 months.
  Interventions: Device: Active video games; Other: tennis training process
- NO-AVI (Active Comparator): The NO_AVI group were involved in a regular tennis training process, two times a week for one hour. The training process lasted 6 months.
  Interventions: Other: tennis training process

INTERVENTIONS:
Device: Active video games — Participants played the active video game Virtua tennis 4 on a playstation kinect device
  Arms: I-AVI
Other: tennis training process — Participants were involved in a regular tennis training process, performed two times a week for one hour per lesson.

SUMMARY:
Developing movement capabilities and efficiently acquiring and assimilating movement information and knowledge in middle childhood stages is of great importance for performing complex movement structures in later stages of life. Our study is directed to researching the influence of active video games (AVG) on assessment of tennis motor skills and visual capabilities in middle childhood, as a part of two separate sub-researches.

DETAILED DESCRIPTION:
In the first sub-research, which included a sample of 55 children aged between 7 and 9, the investigators measured the physiological responses of bodies after acute and chronic exposure to playing AVG. The investigators established a significant difference in skin conductance before beginning the intervention between the virtual and actual game. After the intervention, the experimental group had a significantly higher average value of heart rate frequency and breathing frequency while playing AVG in comparison to the control group.

In the second sub-research the investigators measured progress in tennis technique (TRSC test), development of gross motor skills and change in reaction time on the same group of children. In the TRSC test, the control group improved in all sub-groups with both strokes. The experimental group made no improvements in sub-group 3d with the ''forehand'', 1d and 3d with the ''backhand''. In the gross motor skill development test the investigators have not established a significant interaction effect. In the analogue reaction time measurement test, the investigators recorded a significant interaction between time x group. The same goes for Simon's test with incongruent stimuli, with congruent the interaction was of no relevance.

The investigators established that the use of AVG can represent a new strategy for combining movement/sports activities and cognitively directed tasks aiming at effective assessment of tennis skills.

ELIGIBILITY:
Inclusion Criteria:

* Age limit

Exclusion Criteria:

* excluded were players with injuries or long-term body impairments that prevented them from performing shots as they are usually instructed.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Psychophysiological body responses 1: skin conductance | change from baseline to 3-months intervention
  Skin conductance measured in micro siemens
Psychophysiological body responses 2: skin temperature | change from baseline to 3-months intervention
  Skin temperature measured in Celsius
Psychophysiological body responses 3: heart rate frequency | change from baseline to 3-months intervention
  hear rate measured in beats per minute
Psychophysiological body responses 4: breathing frequency | change from baseline to 3-months intervention
  breathing frequency measured in breaths per minute

SECONDARY OUTCOMES:
TGMD-3 scale (Test of Gross Motor Development-Third Edition) | change from baseline to 3-months intervention
  The TGMD-3 has two subtests. The first subtest, Locomotor, measures the gross motor skills that require fluid coordinated movements of the body as the child moves in one direction or another. The second subtest, Ball Skills, measure the gross motor skills that demonstrate efficient throwing, striking, and catching movements. The TGMD-3 provides an overall composite score (Gross Motor). The two subtest scaled scores are combined to form the Gross Motor composite. The Examiner's Manual discusses the test's theoretical and research-based foundation, item development, standardization, administration and scoring procedures, normative tables, and guidelines for using and interpreting the test's results. The TGMD-3 scale is used to measure the fundamental motor skills in 3-10 year-old children with typical development. The raw score for locomotor subtest is between 0 and 46, while the raw score for ball skills is between 0 and 54. The overall raw score for the test is between 0 and 100.

OTHER OUTCOMES:
Manual/analog visuomotor reaction time task | change from baseline to 3-months intervention
  The time needed to catch a suspended vertical shaft by hand closure, measured in centimeters and then calculated in milliseconds.
Simon task | change from baseline to 3-months intervention
  Congruent and incongruent stimuli measured in milliseconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Tenis klub San Simon Izola, Izola, Slovenia

REFERENCES:
- [Derived] Slosar L, de Bruin ED, Fontes EB, Plevnik M, Pisot R, Simunic B, Marusic U. Additional Exergames to Regular Tennis Training Improves Cognitive-Motor Functions of Children but May Temporarily Affect Tennis Technique: A Single-Blind Randomized Controlled Trial. Front Psychol. 2021 Mar 15;12:611382. doi: 10.3389/fpsyg.2021.611382. eCollection 2021. PMID 33790833